CLINICAL TRIAL: NCT06850662
Title: The Effect of Backward Walking Observation Training on Improving Brain Activity and Gait Quality in People With Stroke
Brief Title: Backward Walking Observation Training in People With Stroke and Gait Quality in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU113210AF2
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Backward walking; Action observation training; Gait symmetry; Gait variability; Brain activity; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Backward walking observation training group (Experimental): The intervention is a 50-minute session and 3 sessions/week, totaling 4 weeks.
  Interventions: Other: Backward walking observation training
- Non-motor observational backward walking training group (Active Comparator): The intervention is a 50-minute session and 3 sessions/week, totaling 4 weeks.
  Interventions: Other: Non-motor observational backward walking training

INTERVENTIONS:
Other: Backward walking observation training — Backward treadmill training after watching a video of backward walking.
  Arms: Backward walking observation training group
Other: Non-motor observational backward walking training — Backward treadmill training after watching a video of landscape without any movements.
  Arms: Non-motor observational backward walking training group

SUMMARY:
Walking impairment is one of the most common and concerning issues for individuals with stroke. Previous studies have often used improvements in walking speed and distance as reference indicators for gait performance progress in individuals with stroke. However, for people with chronic stroke, it may be more appropriate to prioritize improving gait symmetry and gait variability to enhance gait quality as a primary intervention goal. Additionally, stroke can lead to an imbalance in interhemispheric brain activity, which evolves as motor function recovers. According to the literature review, backward walking may extend the support time of the lower limbs, thereby enhancing the weight-bearing capacity of the affected limb. This, in turn, could promote gait symmetry and reduce gait variability. Changes in brain activity might also accompany such improvements in gait quality. Therefore, this study aims to investigate the immediate, short-term and post carryover intervention effects of backward walking observation training on gait quality in individuals with chronic stroke as well as to explore its effects on interhemispheric activity balance in individuals with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 months after the diagnosis of stroke
* Independent walking over at least 7m with or without a walking aid
* Mini-mental state examination score ≥ 24

Exclusion Criteria:

* Had difficulty in backward walking
* Any neuromuscular disorders history
* With visual or auditory disorders
* Unstable cardiac status or uncontrolled hypertension
* Any musculoskeletal disorders that would affect walking ability

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Brain activity | Baseline, 4 weeks after training, and 4-week follow-up
  Using functional near infrared spectroscopy to measure the oxygenated hemoglobin (HbO) and deoxygenated hemoglobin (HbR) in the bilateral prefrontal cortex, supplementary motor area and primary motor cortex.
Gait symmetry | Baseline, post-intervention, 4 weeks after training, and 4-week follow-up
  Using GAITRite system to measure the symmetry of spatiotemporal parameters
Gait varability | Baseline, post-intervention, 4 weeks after training, and 4-week follow-up
  Using GAITRite system to measure the coefficient of variation of spatiotemporal parameters

SECONDARY OUTCOMES:
Gait performance | Baseline, post-intervention, 4 weeks after training, and 4-week follow-up
  Using GAITRite system to measure the gait spatiotemporal parameters
Time Up & Go test | Baseline, 4 weeks after training, and 4-week follow-up
  Using Time Up & Go test to assess functional mobility
Activities-specific Balance Confidence Scale | Baseline, 4 weeks after training, and 4-week follow-up
  Using Activities-specific Balance Confidence Scale to evaluate individual's balance confidence in performing daily activities
Taiwan Chinese version Falls Efficacy Scale | Baseline, 4 weeks after training, and 4-week follow-up
  Using Taiwan Chinese version Falls Efficacy Scale to evaluate concerns about falling

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan